CLINICAL TRIAL: NCT02335970
Title: Effects of a Training Intervention After Thoracoabdominal Oesophagus Surgery -a Randomized Controlled Trial
Brief Title: Effects of a Training Intervention After Thoracoabdominal Oesophagus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FoU in Sweden 13891
Record Dates: First submitted 2014-12-30; First posted 2015-01-12 (Estimated); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Oesophagus Cancer
Keywords: Pain; Range of motion; Quality of life
MeSH Terms: conditions — Esophageal Neoplasms; Pain | interventions — Sensitivity Training Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training group (Experimental): Training program: Daily exercises for 3 months
  Interventions: Other: Training group
- Controls (No Intervention): Standard care

INTERVENTIONS:
Other: Training group — After 1 week
  * Chest expansions
  * Static thoracic extension in prone
  * Lateral flexion of the spine in standing
  * Bilateral shoulder flexion
  * Shoulder external rotation of shoulders
  * Rotation of the thoracic spine in sitting
  * Static back extensor strength in prone
  After 1 month
  * Thoracic extension, rotation and flexion abduction
  * Hand in neck and in back
  * Bilateral active flexion abduction
  * Strength training of leg muscles
  * Static back extensor strength
  After 2 months
  * Strength training of legs and back muscles
  * Push-ups against a wall
  * Thoracic extension in sitting and standing
  * Thoracic rotation in lying
  * Stretching of mm. pectoralis Training was performed daily with 10 rep of each exercise
  Arms: Training group

SUMMARY:
This study evaluates the effect of a training intervention after thoracoabdominal resection of the oesophagus. Half of the patients scheduled for thoracoabdominal oesophagus surgery were randomized to an intervention group while the other half a control group.

DETAILED DESCRIPTION:
It is well known that thoracoabdominal oesophageal resection for cancer is a procedure with high risks for complications. Earlier trials have shown that respiratory restrictions persist after the operation as well as lower physical function, range of motion in the rib-cage and limitations in activities in daily living. There are, however, only two clinical studies that evaluate postoperative breathing exercises and none evaluating any other rehabilitation interventions.

In other types of extensive surgery that may affect mobility with trauma to muscles and bone structures in the thorax and thoracic spinal column, there is strong evidence that speaks for an active rehabilitation approach in favour of a less active one.

The intervention evaluated was a rehabilitation program including exercises to restore lung function, range of motion in the thoracic spine and shoulders and strength exercises for the back extensors, shoulders and legs.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for thoracoabdominal oesophageal resection
* Ability to perform 90 W during a sub-maximal bicycle test
* Ability to speak Swedish

Exclusion Criteria:

* Serious untreated cardiac disease that may be critical
* Musculoskeletal or neurological disease or trauma affecting respiration or range of motion in the rib cage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2005-09-05 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Degree of physical disability estimated by the Disability Rating Index (DRI) | 3 months
  12 items covering activities from dressing and going for walks to lifting heavy objects and exercising. The item responses were rated on visual analogue scales (0-100)

SECONDARY OUTCOMES:
Pain in the neck, rib cage and shoulders (visual analogue scale) | 3 months
  Estimated on a 100-mm visual analogue scale
FVC (Forced Vital Capacity) | 3 months
  Forced Vital Capacity performed in a standardised manner
Range of motion | 3 months
  Thorax expansion, back flexion, extension and lateral flexion, shoulder flexion and abduction
Physical function (Time stand test and heel rise test) | 3 months
  Time stand test and heel rise test
Physical Activity (six-level scale) | 3 months
  A six-level scale where low figures indicate a sedentary and a high score an active lifestyle according to Grimby et al
Quality of Life by EORTC QLQ-C30 | 3 months
  European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core -30 version 3.0. All responses were converted to a score of between 0 and 100 using a linear transformation following EORTC guidelines (EORTC). High scores indicate good functioning but a high level of symptoms
FEV1 s | 3 months
  Forced performed in a standardised manner
PEF (Peak Expiratory Flow) | 3 months
  Peak Expiratory Flow performed in a standardised manner

CONTACTS AND LOCATIONS:
Overall Officials: Monika Fagevik Olsén, PhD, Principal Investigator — Professor at Sahlgrenska Academy at Gothenburg University, Sweden